CLINICAL TRIAL: NCT03499730
Title: Does Preoperative Midazolam Dose Affect Postoperative Pain? - a Multicentric Observational Study in Open Inguinal Hernia Repair
Brief Title: Does Midazolam Affect Postoperative Pain?
Status: Completed | Type: Observational
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, Caroline Dahlem, Principal Investigator, Universidade do Porto
Other Study IDs: Midazolam OBS
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Pain, Postoperative
Keywords: Midazolam; Inguinal hernia
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal | interventions — Midazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Midazolam injection — The dose of preoperative midazolam is the predictor variable and will be registered as a continuous variable in a single cohort.

SUMMARY:
To investigate whether midazolam has any effect on postoperative pain in outpatient surgery, the investigators will assess the impact of different midazolam doses on pain scores 24h, 7 days and 3 months after open inguinal hernia repair.

The investigators hypothesize that patients being administered higher midazolam doses will refer more pain.

DETAILED DESCRIPTION:
Systemic midazolam prescribed perioperatively might have impact on pain, with studies suggesting antinociceptive and hyperalgesic effects. Anxiety might be a confounder in this association. In order to investigate the effect of midazolam on postoperative pain, a prospective cohort study will be conducted in four Portuguese ambulatory surgery units. A convenience sample with consecutive design will include patients admitted for open inguinal hernia repair. After anxiety and pain evaluation, a tailored dose of midazolam will be administered as premedication according to the anesthetist's best judgement within each unit's protocol (routine care; this dose may be null). Subsequent anesthesia and analgesia will be standardized. Postoperative pain will be blindly assessed by telephone interviews at 24h, 7 days, and 3 months. Statistical analysis will be performed separately for each gender, centre and type of anesthesia, adjusting for preoperative anxiety and other confounding variables with multivariate analysis.

The investigators intend to clarify the relation between anxiety, preoperative midazolam and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

- adults proposed for open inguinal hernia repair in Portuguese ambulatory surgery units

Exclusion Criteria:

* psychiatric disorders
* alcoholism
* illiteracy or poor understanding of the Portuguese language
* history of chronic pain under opioids
* recurrent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients proposed for open inguinal hernia repair in Portuguese ambulatory surgery units, under general or spinal anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 24h after surgery
  Pain numeric rating scale (NRS) 0-10

SECONDARY OUTCOMES:
Postoperative pain | 7 days after surgery
  Pain NRS
Postoperative pain | 3 months after surgery
  Pain NRS
Patient satisfaction | 7 days after surgery
  NRS
Patient satisfaction | 3 months after surgery
  NRS
Analgesic consumption | 24h after surgery
  Total analgesic drugs taken in a time period
Analgesic consumption | 7 days after surgery
  Total analgesic drugs taken in a time period
Adverse events | 7 days after surgery
  Number of patients with adverse events like bleeding, nausea, uncontrolled pain
Global surgery recovery index | 3 months after surgery
  Global surgery recovery index

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Dahlem, MD, Principal Investigator — UPorto /CINTESIS
Locations (4):
- Portugal (4):
  - Centro Hospitalar Baixo Vouga, EPE, Aveiro
  - Centro Hospitalar Universitário do Algarve, Faro
  - Centro Hospitalar Entre Douro e Vouga, EPE, Santa Maria da Feira
  - Centro Hospitalar Vila Nova de Gaia / Espinho, EPE, Vila Nova de Gaia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article might be shared with other researchers after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 6 months following article publication.
Access Criteria: Proposals should be directed to caroline.dahlem@gmail.com. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Mantegazza P, Parenti M, Tammiso R, Vita P, Zambotti F, Zonta N. Modification of the antinociceptive effect of morphine by centrally administered diazepam and midazolam. Br J Pharmacol. 1982 Apr;75(4):569-72. doi: 10.1111/j.1476-5381.1982.tb09175.x. PMID 6121598
- [Background] Okulicz-Kozaryn I, Kaminska E, Luczak J, Szczawinska K, Kotlinska-Lemieszek A, Baczyk E, Mikolajczak P. The effects of midazolam and morphine on analgesic and sedative activity of ketamine in rats. J Basic Clin Physiol Pharmacol. 2000;11(2):109-25. doi: 10.1515/jbcpp.2000.11.2.109. PMID 11037766
- [Background] Tatsuo MA, Salgado JV, Yokoro CM, Duarte ID, Francischi JN. Midazolam-induced hyperalgesia in rats: modulation via GABA(A) receptors at supraspinal level. Eur J Pharmacol. 1999 Apr 1;370(1):9-15. doi: 10.1016/s0014-2999(99)00096-5. PMID 10323274
- [Background] Frolich MA, Zhang K, Ness TJ. Effect of sedation on pain perception. Anesthesiology. 2013 Mar;118(3):611-21. doi: 10.1097/ALN.0b013e318281592d. PMID 23314164
- [Background] Kain ZN, Sevarino F, Pincus S, Alexander GM, Wang SM, Ayoub C, Kosarussavadi B. Attenuation of the preoperative stress response with midazolam: effects on postoperative outcomes. Anesthesiology. 2000 Jul;93(1):141-7. doi: 10.1097/00000542-200007000-00024. PMID 10861157
- [Background] Coulthard P, Rood JP. An investigation of the effect of midazolam on the pain experience. Br J Oral Maxillofac Surg. 1992 Aug;30(4):248-51. doi: 10.1016/0266-4356(92)90268-n. PMID 1510899
- [Background] Day MA, Rich MA, Thorn BE, Berbaum ML, Mangieri EA. A placebo-controlled trial of midazolam as an adjunct to morphine patient-controlled analgesia after spinal surgery. J Clin Anesth. 2014 Jun;26(4):300-8. doi: 10.1016/j.jclinane.2013.12.011. Epub 2014 Jun 2. PMID 24882605
- [Background] Hasani A, Maloku H, Sallahu F, Gashi V, Ozgen SU. Preemptive analgesia with midazolam and diclofenac for hernia repair pain. Hernia. 2011 Jun;15(3):267-72. doi: 10.1007/s10029-010-0772-y. Epub 2010 Dec 28. PMID 21188440
- [Background] Ong CK, Seymour RA, Tan JM. Sedation with midazolam leads to reduced pain after dental surgery. Anesth Analg. 2004 May;98(5):1289-93, table of contents. doi: 10.1213/01.ane.0000111107.18755.cc. PMID 15105203